CLINICAL TRIAL: NCT02787109
Title: A Phase I First in Human, Double-blind, Parallel, Randomised and Placebo Controlled Clinical Trial of the Safety of SSI's Adjuvanted Chlamydia Vaccine CTH522 in Healthy Women Aged 18 to 45 Years
Brief Title: Safety of Chlamydia Vaccine CTH522 in Healthy Women Aged 18 to 45 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHLM-01
Record Dates: First submitted 2016-05-23; First posted 2016-06-01 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Chlamydia Trachomatis
Keywords: Safety; Immunogenicity; Phase I

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CTH522-CAF01 (Experimental): CTH522-CAF01: CTH522 chlamydia antigen adjuvanted with CAF01 for IM administration (preferably the non-dominant arm)
  CTH522 chlamydia antigen diluted with Tris buffer for IN administration
  Interventions: Biological: CTH522-CAF01
- CTH522-Al(OH)3 (Experimental): CTH522-Al(OH)3: CTH522 chlamydia antigen adjuvanted with aluminium hydroxide, Al(OH)3 , for IM administration (preferably the non-dominant arm)
  CTH522 chlamydia antigen diluted with Tris buffer for IN administration
  Interventions: Biological: CTH522-Al(OH)3
- Placebo (Placebo Comparator): Saline for IM and In administrations
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CTH522-CAF01 — CTH522 chlamydia antigen adjuvanted with CAF01 for IM administration
  Arms: CTH522-CAF01
Biological: CTH522-Al(OH)3 — CTH522 chlamydia antigen adjuvanted with aluminium hydroxide, Al(OH)3 , for IM administration
  Arms: CTH522-Al(OH)3
Biological: Placebo — Saline
  Arms: Placebo

SUMMARY:
The present trial is a phase I first in human, double blind, parallel and placebo controlled trial of SSI's adjuvanted chlamydia vaccine CTH522: CTH522-CAF01 (CAF01 is an adjuvant system) and CTH522-Al(OH)3. The trial will be conducted at Imperial College Research site in the United Kingdom.

Subjects are randomly assigned to one of the following three treatment groups in a ratio of 3:3:1.

This trial consisted of 10 visits and 5 telephonic interviews

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy female between 18 and 45 years of age on the day of first trial vaccination
2. Has provided signed informed consent
3. Is willing and likely to comply with the trial procedures
4. Is prepared to grant authorised persons access to their medical record
5. Willing to use acceptable contraceptive measures* during the trial (2 weeks before and 2 weeks after the trial)

   * Heterosexually active female capable of becoming pregnant must (in addition to requiring male partner to use condoms) agree to use hormonal contraception, or to complete abstinence, from at least 2 weeks before the first vaccination until at least 2 weeks after the last. (Note: Periodic abstinence [e.g. calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal and intrauterine device or intrauterine hormone releasing system and progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action, are not acceptable methods of contraception)

Exclusion Criteria:

1. Has confirmed history of Pelvic Inflammatory Disease or significant gynaecological diseases
2. Is positive for C. trachomatis (PCR)
3. Is positive for gonorrhoea (urine), HIV, Hepatitis B/C, syphilis (blood)
4. Has a positive pregnancy test
5. Has a significant active disease - such as cardiac, liver, immunological, neurological, psychiatric; or clinically significant abnormality of haematological or biochemical parameters.
6. Has BMI of 35 kg/m2 or greater
7. Is currently participating in another clinical trial with an investigational or noninvestigational drug or device
8. Has received, or plans to receive, an active immunisation within 14 days of the start of the trial or any of the immunisation visits in this trial
9. Is currently receiving treatment with immunosuppressive agents e.g. oral, inhaled, nasal or injected corticosteroids. (Topical steroids are allowed, unless applied to the IM injection site.)
10. Is using an intrauterine device
11. Has a condition which in the opinion of the investigator is not suitable for participation in the trial
12. Known or confirmed allergy to any of the vaccine constituents -

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2016-07; Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of adverse events/reactions and laboratory safety of adjuvanted chlamydia vaccine | Through study completion (Day 0 to Day 168)
  Solicited local injection site reactions (recorded at any visit) after intramuscular (IM) administration (pain, erythema, tenderness, pruritus, warmth, stiffness and swelling) Solicited local reactions (recorded at any visit) after IN administration (discharge, including bleeding, congestion, discomfort, sneezing and cough) Solicited systemic reactions (recorded at any visit) after IM and IN administration (abnormally raised temperature, chills, myalgia, malaise, fatigue, rash, headache, nausea and vomiting, and clinically significant abnormal values among full blood count, liver function test and renal profile results)

SECONDARY OUTCOMES:
Serum immunoglobulin G antibody responses after vaccination with CTH522 | At Days 0, 28, 112, 126, 140, 154 and 168
  Percentage of subjects achieving seroconversion for anti-CTH522 immunoglobulin G antibody at any time points after IM vaccination(s)

CONTACTS AND LOCATIONS:
Overall Officials: Sonya Abraham, Principal Investigator — Imperial College London
Locations (1):
- NIHR/Wellcome Trust Imperial Clinical Research Facility, Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abraham S, Juel HB, Bang P, Cheeseman HM, Dohn RB, Cole T, Kristiansen MP, Korsholm KS, Lewis D, Olsen AW, McFarlane LR, Day S, Knudsen S, Moen K, Ruhwald M, Kromann I, Andersen P, Shattock RJ, Follmann F. Safety and immunogenicity of the chlamydia vaccine candidate CTH522 adjuvanted with CAF01 liposomes or aluminium hydroxide: a first-in-human, randomised, double-blind, placebo-controlled, phase 1 trial. Lancet Infect Dis. 2019 Oct;19(10):1091-1100. doi: 10.1016/S1473-3099(19)30279-8. Epub 2019 Aug 12. PMID 31416692